CLINICAL TRIAL: NCT05174845
Title: An Observational, Retrospective and Multicenter Study to Evaluate the Effectiveness and Safety of 1L (PEG)+ Ascorbic Acid Given for Bowel Preparation Prior to Colonoscopy in Iberia
Brief Title: Real Word Evidence With 1L Polyethylene Glycol (PEG)+ Ascorbic Acid in Iberia
Status: Completed | Type: Observational
Sponsor: Norgine (Industry)
Collaborators: Xolomon Tree S.L. (Unknown)
Responsible Party: Sponsor
Other Study IDs: PLEN-01/2021
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Colon Cancer; Colon Disease; Colon Cleansing
MeSH Terms: conditions — Colonic Neoplasms; Colonic Diseases | interventions — Ascorbic Acid; Polyethylene Glycols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: 1L PEG + ASCORBIC ACID — * 2-Day Split-Dosing: The patient has taken the product in the evening before the scheduled colonoscopy and mandatory additional clear fluid. The patient has taken the second dose with mandatory additional clear fluids on the morning of the colonoscopy.
  * Same Day: The patient has taken the first dose of the product on the day of the colonoscopy and take mandatory additional clear fluid. After a 1-2 hour break, the patient has taken a second dose plus additional clear mandatory fluid.
  Other Names: PLENVU; NER1006; PLEINVUE

SUMMARY:
A retrospective study to evaluate the effectiveness and safety of 1L polyethylene glycol (PEG)+ Ascorbic acid given for bowel preparation before colonoscopy.

DETAILED DESCRIPTION:
Observational, retrospective, and multicenter study based on the review of the existing medical records of patients followed on an outpatient basis (computerized databases and dissociated data).

The design implies the incorporation of existing anonymized data by the hospital centers without leaving any record of the code assigned to each patient. The design, therefore, avoids the possible risk of the dissemination of the personal data of patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients aged: ≥18 years undergoing a screening, surveillance, or diagnostic colonoscopy between June 1, 2019, to September 1, 2021
* Who have used NER1006 in the preparation of the colonoscopy either in split doses or same day.

Exclusion Criteria:

* History of colorectal cancer o colectomy before the first colonoscopy
* Impossibility to obtain the required mandatory data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All outpatients aged: ≥18 years undergoing a screening, surveillance, or diagnostic colonoscopy who have prepared with NER1006
Sampling Method: Non-Probability Sample
Enrollment: 13393 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Number of patients With Successful Bowel Cleansing (Overall Colon) | Up to 2 days (from day of first dosing to day of colonoscopy)
  The proportion of patients with adequate total colon cleansing is defined as a Boston Bowel preparation scale (BBPS) score ≥ 2 in all segments (BBPS> 6).
Number of Patients With 'Excellent Plus Good' (Highly Effective) Bowel Cleansing (Colon Ascendens) | Up to 2 days (from day of first dosing to day of colonoscopy)
  Proportion of patients with a high-quality cleaning in the right colon defined as a BBPS score = 3.

SECONDARY OUTCOMES:
Polyps Detection Rate in the total colon and in the right colon | Up to 2 days (from day of first dosing to day of colonoscopy)
  Proportion of colonoscopies where at least one polyp was found and removed in total and right colon
Adenoma Detection Rate in the total colon and in the right colon | Up to 2 days (from day of first dosing to day of colonoscopy)
  Proportion of colonoscopies where at least one adenoma is found based on histological analysis in total and right colon
Cecal intubation rate | Up to 2 days (from day of first dosing to day of colonoscopy)
  Defined as the visualization of the ileocecal valve and / or appendicular orifice
Cecal intubation time | Up to 2 days (from day of first dosing to day of colonoscopy)
  Defined as the time required for the introduction of the colonoscope to reach the base of the cecum.
Withdrawal time | Up to 2 days (from day of first dosing to day of colonoscopy)
  Defined as the minutes spent inspecting the colon wall.
Tolerability of the preparation, if available | Up to 2 days (from day of first dosing to day of colonoscopy)
  Defined as good, fair or poor.
Tolerability of the preparation, if available | Up to 2 days (from day of first dosing to day of colonoscopy)
  Defined with a semi-quantitative scale of 1-5 (1 = totally agree, 2 = agree, 3 = Neutral, 4 = disagree, 5 = totally disagree)
Adherence to the preparation, if available. | Up to 2 days (from day of first dosing to day of colonoscopy)
  Percentage of patients with adherence to the preparation, defined as ingestion of at least 75% of each of the two doses
Treatment satisfaction, if available | Up to 2 days (from day of first dosing to day of colonoscopy)
  Percentage of patients satisfied with the preparation
Quality of the preparation (BBPS> 2 in all colon segments) depending on the dietary guideline | Up to 2 days (from day of first dosing to day of colonoscopy)
  Quality of the preparation (BBPS> 2 in all colon segments) depending on the dietary guideline
Safety of the preparation | Up to 2 days (from day of first dosing to day of colonoscopy)
  Safety from registered adverse effects.
Sub-analyzes will be conducted in different patient populations | Up to 2 days (from day of first dosing to day of colonoscopy)
  Patients ≥ 65 years, patients with chronic constipation, with diabetes mellitus, with hypertension, with mild to moderate renal failure and with inflammatory bowel disease.
Sub-analyzes of the primary and secondary outcomes | Up to 2 days (from day of first dosing to day of colonoscopy)
  Sub-analyzes will be carried out by country, by the reason for the colonoscopy and by the recommended dietary regimen

CONTACTS AND LOCATIONS:
Overall Officials: Jose Miguel Esteban López-Jamar, MD, Principal Investigator — Norgine Spain
Locations (12):
- Portugal (2):
  - Hospital da Senhora da Oliveira, Guimarães
  - Hospital CUF Descobertas, Lisbon
- Spain (10):
  - Consorci Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital San Rafael, A Coruña
  - HM Sant Jordi, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Doctor López Cano, Cadiz
  - Complejo hospitalario Ruber Juan Bravo, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital La Zarzuela, Madrid
  - Hospital Quirón salud Sagrado Corazón, Seville
  - Consorcio Hospitalario Provincial de Castelló, Valencia